CLINICAL TRIAL: NCT06618183
Title: User Performance Evaluation of the Intelligent Fingerprinting Drug Screening System: Method Comparison and Usability
Brief Title: Drug Screening System Method Comparison
Status: Recruiting | Type: Observational
Sponsor: Intelligent Bio Solutions Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IBS-2024-02
Record Dates: First submitted 2024-08-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Reagent Kits, Diagnostic
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- 1: Donors randomized into the 0 mg codeine dosage block
  Interventions: Diagnostic Test: Fingerprint sweat drug screen; Diagnostic Test: Fingerprint sweat laboratory analysis
- 2: Donors randomized into the 30 mg codeine dosage block
  Interventions: Diagnostic Test: Fingerprint sweat drug screen; Diagnostic Test: Fingerprint sweat laboratory analysis
- 3: Donors randomized into the 60 mg codeine dosage block
  Interventions: Diagnostic Test: Fingerprint sweat drug screen; Diagnostic Test: Fingerprint sweat laboratory analysis

INTERVENTIONS:
Diagnostic Test: Fingerprint sweat drug screen — Qualitative lateral-flow immunoassay analysis of fingerprint sweat specimen
Diagnostic Test: Fingerprint sweat laboratory analysis — Laboratory analysis of fingerprint sweat specimen by liquid chromatography/tandem mass spectrometry

SUMMARY:
Prospective, open-label, single-dose, randomized, multi-site performance evaluation of the accuracy and usability Intelligent Fingerprinting Drug Screening System in the hands of intended users: "operators" and "donors."

DETAILED DESCRIPTION:
This study will compare positive and negative test results obtained from fingerprint sweat using the Intelligent Fingerprinting DSC-7 Drug Screening Cartridge versus opiates in sweat collected via the Fingerprint Collection Kit for Laboratory Analysis, within healthy males and non-pregnant females.

The primary objective is to compare the sensitivity, specificity, and accuracy of the Intelligent Fingerprinting Drug Screening System to the validated confirmatory LC-MS/MS technique.

The secondary objectives are to assess drug screening system usability and reproducibility.

"Operators" comprise nine (9) adults: male and female subjects who operate the drug screening system. These subjects are not administered any drug. "Operators" represent end users who utilize the screening system in a laboratory setting. "Operators" will be provided the Intelligent Fingerprinting Drug Screening Guide, Confirmatory Laboratory Analysis Guide, and Quick Reference Guide, and be trained in system use. After receiving and reviewing all materials, the "operator" will complete a Training Exam to determine if he or she may proceed with testing.

"Donors" comprise 135 healthy adults: male and non-pregnant female subjects who provide fingerprint sweat specimens. Subjects will be randomized into the blocks administered 0, 30, or 60mg of codeine sulfate in tablet form. "Donors" represent end users either applying for employment or working at an organization that conducts pre-employment and/or periodic workplace drug screening.

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the nature of the study, agreed to, and able to read, review, and sign the informed consent document prior to dosing. The informed consent document will be written in English; therefore, the subject must have the ability to read and communicate in English.
2. *Completed the screening process within 30 days prior to dosing. Subjects screened as a part of an IRB-approved General Screening Protocol at the clinical research site may be included in this study without additional screening procedures, provided all the required screening procedures have been performed within 30 days prior to dosing.
3. Healthy male and non-pregnant female subjects from ages 18 to 65, inclusive, at the time of dosing.
4. *Body mass index (BMI) from 18 kg/m2 to 30 kg/m2, inclusive, and weigh at least 60 kg.
5. *Females of childbearing potential must be willing to practice an acceptable form of contraception (see Section 9.3.3), and have a negative urine pregnancy test on admission to the treatment phase of the study.
6. *Males must agree to practice an acceptable form of contraception.
7. *Judged by the Investigator and/or designee to be in good health as documented by the medical history, and vital sign assessments. Any abnormalities or deviations outside the normal range for vital signs can be repeated by clinical staff and judged to be not clinically significant for study participation.

Exclusion Criteria:

1. Unwilling or unable to provide informed consent.
2. *More than three digits absent from the hands due to congenital or accidental cause(s).
3. *Reports receiving any investigational drug within 30 days prior to dosing.
4. *Reports a clinically significant illness during the 30 days prior to the in-clinic portion of the study (as determined by the Investigator).
5. *Reports any personal history of substance abuse (including drug/alcohol abuse or addiction) or mental illness (e.g. major depression) within one year prior to screening visit.
6. *Is pregnant (females only).
7. *Presence of any clinically significant results from laboratory tests and vital signs assessments, as judged by the Investigator.
8. *Reports history of respiratory depression (e.g., sleep apnea).
9. *Current severe hypotension (i.e., systolic blood pressure <90 mmHg).
10. *Reports known or suspected gastrointestinal obstruction including, paralytic ileus.
11. *Reports current presence of acute bronchial asthma/ upper airway obstruction.
12. *Reports a history of clinically significant allergies, including food or drug allergies, as judged by the Investigator.
13. *Reports history or current condition of adrenal insufficiency.
14. *Reports history or current condition of renal disease.
15. If, in the opinion of the Investigator, the subject is not suitable for the study.

    * Required only for "donors." Not required for "operators."

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, Female
Study Population: Subjects will be recruited from the community at large.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Method Comparison | 30 minutes to 3 hours
  Comparison of the sensitivity, specificity, and accuracy of the Intelligent Fingerprinting Drug Screening System (qualitative lateral-flow immunoassay) to the validated confirmatory LC-MS/MS technique

SECONDARY OUTCOMES:
Usability | 72 hours
  Usability of the Intelligent Fingerprinting Drug Screening System based on scores obtained by operators on written training exam (Drug Screening Process and Laboratory Process Exam). Training exam score must meet or exceed 85% for each operator.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - CenExel iResearch, Decatur, Georgia
  - CenExel HRI, Berlin, New Jersey
  - CenExel HRI, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No